

General Consent Form Template Version Date: January 2019

Protocol Title: Assessing efficacy of IV acetaminophen for perioperative pain control for oocyte retrieval: a randomized, double blind, placebocontrolled trial

Principal Investigator: John C. Petrozza, MD

Site Principal Investigator:

Description of Subject Population: Adult patients undergoing oocyte retrievals under concious sedation

#### **About this consent form**

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

Partners HealthCare System is made up of Partners hospitals, health care providers, and researchers. In the rest of this consent form, we refer to the Partners system simply as "Partners."

If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

## **Key Information**

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. Your decision won't change the medical care you get within Partners now or in the future.

The following key information is to help you decide whether or not to take part in this research study. We have included more details about the research in the Detailed Information section that follows the key information.

## Why is this research study being done?




In this research study we want to learn more about how effective acetaminophen (Tylenol) is at reducing pain and the time in the recovery room after oocyte (egg) retrieval. We will compare three types of pre-operative medications: intravenous (IV) acetaminophen, oral (PO) acetaminophen, and placebo (no medication), which is the current typical care. The standard anesthesia care will be provided afterwards. We also want to find out whether pre-operative acetaminophen can reduce a person's need for opioid pain medications (such as morphine) to "rescue" breakthrough pain.

## How long will you take part in this research study?

You will take part in this research study on the day of your oocyte retrieval. We will also call you for a brief follow-up phone call two days after you are discharged home. No additional office visits will be required.

A member of our study staff will review your medical record to collect data regarding your demographic, clinical, IVF cycle, and pregnancy information, which will be kept confidential for your privacy. This may occur up to one year after your procedure. You do not need to do anything for this part of the study.

## What will happen if you take part in this research study?

If you decide to join this research study, the following things will happen:

You must agree to avoid pain medications during the 24 hours prior to your egg retrieval.

We will then assign you by chance (like a coin toss) to one of three study groups for preoperative (prior to egg retrieval) medication:

- -IV acetaminophen plus oral placebo (pill without medicine)
- -IV placebo (liquid without medicine) plus oral acetaminophen
- -IV placebo plus oral placebo

After being given one of the three above sets of medications, standard anesthesia will be administered during the procedure, and any pain will be treated. You, your nurse, the study staff, and your primary fertility physician will not know which study group you are in. The anesthesiologist providing you with anesthesia during your procedure will know the study group you are in to make sure he or she can safely provide you anesthesia care.




## Why might you choose to take part in this study?

We cannot promise any benefits to you from taking part in this research study. However, possible benefits may include reduced pain after surgery, reduced need for opioid medication, and shorter time to discharge after your retrieval. Other women undergoing egg retrievals may benefit in the future from what we learn in this study.

## Why might you choose NOT to take part in this study?

Taking part in this research study has some risks and requirements that you should consider carefully. Important risks and possible discomforts to know about include primarily side effects from acetaminophen use.

A detailed description of side effects, risks, and possible discomforts can be found later in this consent form in the section called "What are the risks and possible discomforts from being in this research study?"

## What other treatments or procedures are available for your condition?

Other available treatments or procedures that are available for post-operative pain management include IV or oral opioids and NSAIDs. Any post-operative pain will be treated appropriately regardless of participation in the study.

# If you have questions or concerns about this research study, whom can you call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

**John C. Petrozza M.D.** is the person in charge of this research study. You can call him at 617-726-8868, available M-F 9-5. You can also contact **Jingping Wang M.D.**, **Ph.D.** at 617-726-2000 M-F 9-5 with questions about this research study.

If you have questions about the scheduling of appointments or study visits, call Dr. Petrozza at 617-726-8868.

If you want to speak with someone **not** directly involved in this research study, please contact the Partners Human Research Committee office. You can call them at 857-282-1900.

You can talk to them about:

| Subject | Identificat | ion |
|---------|-------------|-----|


- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure to take part in, or to continue in the research study

#### **Detailed Information**

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## Why is this research study being done?

In this research study we want to learn more about how effective certain medications are at reducing pain after oocyte (egg) retrieval surgery and how effective they are at reducing the time between the retrieval and discharge from the hospital. We will compare three types of preoperative medications: intravenous (IV) acetaminophen, oral (PO) acetaminophen, and placebo (no medication), which is the current typical care. The placebo looks exactly like the acetaminophen, but contains no acetaminophen. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

The standard anesthesia care will be provided afterwards. We also want to find out whether IV acetaminophen can reduce a person's need for opioid pain medications (such as morphine) to "rescue" breakthrough pain.

Both forms of acetaminophen are currently approved by the U.S. Food and Drug Administration (FDA) for the treatment of pain.

You have been asked to take part in this study because you are scheduled to have oocyte (egg) retrieval. This study will have three research groups. Each group of the study will have approximately 58 subjects. About 174 people will take part in this research study, all at the Massachusetts General Hospital (MGH)

The New England Fertility Society is funding this study.

## Who will take part in this research?




We are asking you to take part in this rsearch study because you are over age 18 and planning to undergo an egg retrieval as a part of your fertility treatment. Approximately 174 patients will participate in this study at MGH. The New England Fertility Society is providing funding for this study.

## What will happen in this research study?

If you decide to join this research study, the following things will happen:

#### **Prior to Egg Retrieval**

You must agree to avoid pain medications like Tylenol or ibuprofen in the 24 hours prior to your procedure.

#### Day of Egg Retrieval

An MGH Research Pharmacist will then randomly assign you to one of three study groups for pre-operative (prior to egg retrieval) medication:

- -IV acetaminophen plus oral placebo (pill without medicine)
- -IV placebo (liquid without medicine) plus oral acetaminophen
- -IV placebo plus oral placebo

You will have a 1 in 3 chance of being assigned to each of the 3 study groups. You and the study doctor cannot choose your study group. The medications are prepared by the MGH Research Pharmacy.

After signing an informed consent with the IVF docter, you will be given one of the three above sets of medications before your egg retrieval in the pre-operative suite. Next, standard anesthesia will be administered during the procedure, and any pain will be treated. Your nurse will record what pain medications you require in the recovery room and how much pain you are in.

You, your nurse, the study staff, and your primary fertility physician will not know which study group you are in. The anesthesiologist providing you with anesthesia during your procedure will know the study group you are in to make sure he or she can safely provide you anesthesia care.

A notation that you are taking part in this research study may be made in your medical record. Information from the research that relates to your general medical care may be included in the record (for example, list of allergies, results of standard blood tests done at the hospital labs).

#### After Egg Retrieval




You will receive a phone call two days after your egg retrieval to ask you about your recovery and any pain medication used at home. This is the last participation from you for the study.

A member of our study staff will also review your medical record to collect data regarding your demographic, non identifying information, as well as your cycle and pregnancy outcomes. This will occur at three instances, occuring at one month, three months, and one year occur up to one year after your procedure.

#### **Stopping the Study Early**

If you decide to stop taking part in the study for any reason, you may do so at any time.

The study doctor may also take you out of the study without your permission.

This may happen because:

- Acetaminophen or other pain medication was used in the 24 hours prior to surgery.
- In the unlikely event that you are unable to participate in the study due to unexpected events such as requiring intubation, surgery, transfusion, or intensive care after your procedure.

## How may we use and share your samples and health information for other research?

Your health information collected for this study will NOT be used or shared for other research, even if we remove identifiable information like your name, medical record number, or date of birth.

## Will you get the results of this research study?

No. The research study we are doing is only a stepping stone in understanding pain management during and after egg retrieval. Therefore, no information about the results of this research study or the results of your individual participation in the research study will be given to you or your doctor.

# What are the risks and possible discomforts from being in this research study?




Important risks and possible discomforts to know about include primarily side effects from acetaminophen use. Any postoperative pain will be treated regardless of study participation or group.

#### Risks of IV and Oral Acetaminophen (Tylenol)

- This study medication contains acetaminophen. It is not safe to take more than 4 grams (4,000 milligrams) total of acetaminophen in one day. For Tylenol® Extra Strength, it is not safe to take more than 3 grams (3,000 milligrams) in one day. In this study, only 1 gram of acetaminophen will be given.
- Other risks include: nausea, vomiting, headache, and insomnia (inability to sleep) in adult patients
- Some of the rare, but serious risks include: anaphylaxis (allergic reaction) or hepatotoxicity (liver damage)

## Call your doctor right away or seek urgent medical attention if you notice any of these side effects post-operatively:

- Rash, swelling in face, difficulty breathing, or any other concerns for allergic reaction
- Blistering, peeling, or red skin rash (IV form)
- Pain, itching, burning, swelling, or a lump under your skin where the needle was placed (IV form)
- Dark urine or pale stools, nausea, vomiting, loss of appetite, severe stomach pain, yellow skin or eyes
- Pain that lasts longer than 5 days

#### **Risks of loss of Confidentiality**

Despite multiple methods to protect patient privacy, breaches in confidentiality are possible. We will have several procedures in place to minimize this.

#### **Unknown Risks**

There may be other risks that are currently unknown.

## What are the possible benefits from being in this research study?

We cannot promise any benefits to you from taking part in this research study. However, possible benefits may include reduced pain after surgery, reduced need for opioid medication, and shorter time to discharge after your retrieval. Other women undergoing egg retrievals may




benefit in the future from what we learn in this study because we may be able to effectively treat their pain with reduced amounts of opioids and discharge them sooner from the recovery room.

## What other treatments or procedures are available for your condition?

Any pain that you experience during or after your egg retrieval procedure will be treated as appropriate. Other treatments for perioperative pain include: IV or PO opioids (fentanyl, morphine, oxycodone, hydromorphone). NSAIDs such as motrin or toradol are also sometimes used for pain control in patients who are not planning to undergo fresh embryo transfer. However, NSAIDs will not be used in study patients post-operatively in the recovery room in order to consistently assess the impact of pre-operative acetaminophen in all study patients regardless of transfer timing. Usual standard of care for management of post-operative pain at home with Tylenol (transfer patients) or Tylenol and NSAIDs (non-transfer patients) will still apply.

# Can you still get medical care within Partners if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within Partners now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

## What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

## Will you be paid to take part in this research study?

You will not be paid for taking part in this research study.




## What will you have to pay for if you take part in this research study?

Study funds will pay for certain study-related items and services. We may bill your health insurer for, among other things, routine items and services you would have received even if you did not take part in the research. You will be responsible for payment of any deductibles and copayments required by your insurer for this routine care or other billed care. If you have any questions about costs to you that may result from taking part in the research, please speak with the study doctors and study staff. If necessary, we will arrange for you to speak with someone in Patient Financial Services about these costs.

# What happens if you are injured as a result of taking part in this research study?

We will offer you the care needed to treat any injury that directly results from taking part in this research study. We reserve the right to bill your insurance company or other third parties, if appropriate, for the care you get for the injury. We will try to have these costs paid for, but you may be responsible for some of them. For example, if the care is billed to your insurer, you will be responsible for payment of any deductibles and co-payments required by your insurer.

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the beginning of this consent form.

## If you take part in this research study, how will we protect your privacy?

Federal law requires Partners to protect the privacy of health information and related information that identifies you. We refer to this information as "identifiable information."

#### In this study, we may collect identifiable information about you from:

- Past, present, and future medical records
- Research procedures, including research office visits, tests, interviews, and questionnaires




## Who may see, use, and share your identifiable information and why they may need to do so:

- Partners researchers and staff involved in this study
- The sponsor(s) of the study, and people or groups it hires to help perform this research or to audit the research
- Other researchers and medical centers that are part of this study
- The Partners ethics board or an ethics board outside Partners that oversees the research
- A group that oversees the data (study information) and safety of this study
- Non-research staff within Partners who need identifiable information to do their jobs, such as for treatment, payment (billing), or hospital operations (such as assessing the quality of care or research)
- People or groups that we hire to do certain work for us, such as data storage companies, accreditors, insurers, and lawyers
- Federal agencies (such as the U.S. Department of Health and Human Services (DHHS) and agencies within DHHS like the Food and Drug Administration, the National Institutes of Health, and the Office for Human Research Protections), state agencies, and foreign government bodies that oversee, evaluate, and audit research, which may include inspection of your records
- Public health and safety authorities, if we learn information that could mean harm to you
  or others (such as to make required reports about communicable diseases or about child
  or elder abuse)

• Other: N/A

Some people or groups who get your identifiable information might not have to follow the same privacy rules that we follow and might use or share your identifiable information without your permission in ways that are not described in this form. For example, we understand that the sponsor of this study may use your identifiable information to perform additional research on various products or conditions, to obtain regulatory approval of its products, to propose new products, and to oversee and improve its products' performance. We share your identifiable information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. The sponsor has agreed that it will not contact you without your permission and will not use or share your identifiable information for any mailing or marketing list. However, once your identifiable information is shared outside Partners, we cannot control all the ways that others use or share it and cannot promise that it will remain private.




Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your identifiable information. Your permission to use and share your identifiable information does not expire.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifiable information **will not** be used for these purposes without your specific permission.

#### **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your identifiable information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your identifiable information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study.

You have the right to see and get a copy of your identifiable information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.

## **Informed Consent and Authorization**

#### **Statement of Person Giving Informed Consent and Authorization**

- I have read this consent form.
- This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study.
- I have had the opportunity to ask questions.
- I understand the information given to me.

#### **Signature of Subject:**

## **Partners HealthCare System Research Consent Form** Subject Identification **General Consent Form Template Version Date: January 2019** I give my consent to take part in this research study and agree to allow my health information to be used and shared as described above. Subject Time (optional) Date **Signature of Study Doctor or Person Obtaining Consent: Statement of Study Doctor or Person Obtaining Consent** • I have explained the research to the study subject. • I have answered all questions about this research study to the best of my ability. Study Doctor or Person Obtaining Consent Time (optional) Date

Consent Form Version: 1
Consent Form Date: 7-31-2019